CLINICAL TRIAL: NCT06079944
Title: Effects of Progressive Resistance Training Combined With Traditional Physical Therapy in Patients With Shoulder Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/18
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Exercises, Impingement syndrome, Physical therapy , Resistance training, Shoulder pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Motor Activity; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A- Control group (Active Comparator): Group (A)/ control group Involves participants receiving
  1. TENS+ hot pack (10mins)
  2. Pendulum exercises and stretching exercises This group will not receive resistance training from 5 repetitions to 20 repetitions of door way stretch (maintained for 30seconds), pendulum exercises and foam roll strtech will be provided over the 6 weeks protocol
  Interventions: Procedure: Traditional physical therapy
- Group B- Study Group (Experimental): Group (B)/ Experimental group involves participants receiving Traditional l physical therapy for shoulder impingement syndrome for 6 weeks.
  1. TENS+ hot pack (10mins)
  2. Pendulum exercises and stretching exercises 3-6RM Load will be determined after which multipulley system will be used for treatment and treatment will be divided in to two series of 8 repetition: 25%, 30%,35%,40%, 50% of 6RM over the period of 6 weeks Speed of movement will be 2 seconds for both the eccentric and concentric phases.
  To strengthen the shoulder muscles patients will perform flexion, extension, medial and lateral rotation It is a combined treatment so study group will receive both study group and control group intervention
  Interventions: Procedure: Progressive resistance training; Procedure: Traditional physical therapy

INTERVENTIONS:
Procedure: Progressive resistance training — * 6RM Load will be determined after which multipulley system will be used for treatment and treatment will be divided in to two series of 8 repetition:
  * 25%, 30%,35%,40%, 50% of 6RM over the period of 6 weeks
  * Speed of movement will be 2 seconds for both the eccentric and concentric phases.
  * To strengthen the shoulder muscles patients will perform flexion, extension, medial and lateral rotation using multipulley system.
  Arms: Group B- Study Group
Procedure: Traditional physical therapy — * TENS+ Hot pack
  * Pendulum exercises and stretching exercises

SUMMARY:
A randomized control trial will be done on diagnosed Shoulder impingemnet patients with physical therapy screening in Fauji Foundation Hospital Rawalpindi.

There is a growing demand on finding treatments which can be more beneficial and can be started early on in the treatment phase, nowadays.

The purpose of the study is to determine the "effects of progressive resistance training combined with traditional physical therapy in patients with shoulder impingement syndrome" using the resistance band and multipulley system.

The traditional physical therapy will include hot pack placed on shoulder and neck region for ten minutes, Transcutaneous electrical nerve stimular will be used and the electrodes will be placed on the desired area (shoulder complex) the intensity will be increased manually according to the capacity of the patient and the treatment time will be of 15 minutes, stretching exercises such as doorway stretch and foam roll supine stretch will be done in the hospital for first 3 weeks and the next 3 weeks will be for home exercises moving from 5 repetitions to 20 repetitions for a set of 3. stretch will be hold for 30 seconds

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To determine the effect of progressive resistance training combined with traditional physical therapy in patients with shoulder impingement syndrome in terms of strength.
2. To determine the effect of progressive resistance training combined with traditional physical therapy in patients with shoulder impingement syndrome in terms of pain.
3. To determine the effect of progressive resistance training combined with traditional physical therapy in patients with shoulder impingement syndrome in terms of range of motion.

1.HYPOTHESIS:

Alternate Hypothesis:

1. There is significant effect in the study group in terms of pain with progressive resistance training than in control group with traditional physical therapy in patients with shoulder impingement syndrome.
2. There is significant effect in the study group in terms of range of motion with progressive resistance training than in the control group with traditional physical therapy in patients with shoulder impingement syndrome.
3. There is significant effect in the study group in terms of strength with progressive resistance training than in the control group with traditional physical therapy in patients with shoulder impingement syndrome.

Null Hypothesis:

1. There is no significant effect in the study group in terms of pain with progressive resistance training than in control group with traditional physical therapy in patients with shoulder impingement syndrome.
2. There is no significant effect in the study group in terms of range of motion with progressive resistance training than in the control group with traditional physical therapy in patients with shoulder impingement syndrome.
3. There is no significant effect in the study group in terms of strength with progressive resistance training than in the control group with traditional physical therapy in patients with shoulder impingement syndrome.

Research Design: Experimental study. Randomized Control Trial

Clinical setting: Rehabilitation department, Fauji Foundation Hospital Study duration: 18 months

Selection Criteria:

Inclusion Criteria Both genders (Male and Female) Young early adulthood with age 20-40 years. Diagnosed Cases of Shoulder impingement syndrome.

Exclusion criteria:

Active joint disease (rheumatoid, or any other rheumatological disease) Any history of Cardiovascular events Recent history of upper limb surgery Hematological disease. Osteoporosis. Osteomyelitis Active fractures/ non or mal-union fractures Rotator cuff tears Adhesive capsulitis. Sampling technique: Convenience sampling envelope Method

Outcome Measures:

1. Data will be collected on Demographics and general information
2. Pain will be assessed with the help of NPRS (numeric pain rating scale Scale)
3. Strength will be measured while calculating the repetition maximum
4. Range of motion will be calculated by Goniometry
5. self rated upper extremity disability will be measured by DASH (disabilities of Arm, shoulder and hand) questionnaire

Study Group (B) = This group will receive TENS+ Hot pack, Pendulum exercises and stretching exercises for first two weeks before moving to the strength training to avoid any damage incase patient is in the inflammatory phase

* 6RM Load will be determined after which resistance band and multipulley system will be used for treatment and treatment will be divided in to a series of 8 repetitions: 25%, 30%, 35%, 40%, and 50% of 6RM over the period of 6 weeks. Speed of movement will be 2 seconds for both the eccentric and concentric phases.
* To strengthen the shoulder muscles patients will perform flexion, extension, medial and lateral rotation using multipulley system.

Resistance training will only be given to the study group. This groups outcome meaures will be assessed at 3 weeks and then 6th week.

Control group (B) =this group will not receive resistance training through resistance band and multipulley, only traditional Physical therapy will be given and their outcomes will be observed at the baseline and then after treatment of 6 weeks.

Data analysis techniques:

Firstly, Informed consent will be taken by the participants. Data will be gathered according to the inclusion criteria mentioned in the study. Screening tests will be applied and if patient reports the following tests positive: Painful Arc Sign, Infraspinatus test, and Hawkin Kennedy then there is a high likelihood ratio of having the disease and if all three tests are negative, there is strong evidence of absence of disease. Tests for other muscles will also be applied that passes through the subacromial space. Pain will be scored using numeric pain rating scale before the assignment of population in both the groups. Convenience sampling will be used to include the participants in either the control group or study group.

Significance of the study:

1. Progressive resistance training program for the musculature of the shoulder in patients with shoulder impingement syndrome may prove effective in reducing pain, increasing strength and improving function.
2. This study will help the practitioner to use the new treatment options for treating patients with shoulder impingement syndrome.
3. The results of the study will add to the literature about the effects of progressive resistance training combined with traditional physical therapy in patients with shoulder impingement syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.(Male and Female)
* Young early adulthood with age 20-40 years.
* Diagnosed cases of Shoulder impingement syndrome.

Exclusion Criteria:

* Active joint disease (rheumatoid, or any other rheumatological diseases
* Any history of Cardiovascular events
* Any history of upper limb surgery
* Hematological disease.
* Osteoporosis.
* osteomyelitis
* Active fractures/ non or mal-union fractures
* Rotator cuff tears
* Adhesive capsulitis.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity using Numeric pain rating scale (NPRS) | 6 weeks
  change in the values of pain using Numeric pain rating scale from the base line then week 3 and then to the end of 6 weeks
Shoulder range of motion using Goniometer | 6 weeks
  Shoulder range of motion will be assessed using goniometer in flexion, extension, abduction, external and internal rotation of shoulder for both the study and control group

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan